CLINICAL TRIAL: NCT04457375
Title: Skin Biophysical Measures for Assessing Head and Neck Cancer-Related External Lymphedema
Status: Completed | Type: Observational
Sponsor: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Harvey Mayrovitz, Professor, Nova Southeastern University
Other Study IDs: 2019-595-NSU
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Lymphedema, Secondary
Keywords: tissue dielectric constant; head and neck lymphedema; lymphedema; reference values
MeSH Terms: conditions — Lymphedema; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Adults: Healthy
  Interventions: Diagnostic Test: TDC

INTERVENTIONS:
Diagnostic Test: TDC — measurements

SUMMARY:
Selected measurements in healthy persons of skin tissue dielectric constant as reference values for subsequent use to evaluate patients with head and neck lymphedema.

DETAILED DESCRIPTION:
Skin tissue dielectric constant (TDC) measurements will non-invasively be made bilaterally at two neck sites, bilaterally on two forearm sites and one site at the chin sub-mental area.

Measurements are made with subjects fully clothed and seated. Measurements are made in triplicate and averaged at each site. Full measurements take about 5-7 minutest to complete. Data will be analyzed to determine the neck-to-arm ratios and chin-to-arm ratios to establish normal ranges of these parameters for subsequent use as comparisons to evaluate and track changes in patients with head and neck lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Healthy with no current or past skin conditions affecting neck or arms

Exclusion Criteria:

1. Known to have diabetes of any type.
2. Having facial or neck hair that prohibits accurate measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Neck-to-Arm TDC ratio | one year
  Neck-to-Arm TDC ratio
Sub-Mental-to-Arm TDC ratio | one year
  Sub-Mental-to-Arm TDC ratio

SECONDARY OUTCOMES:
Bilateral values and Variability in TDC values | one year
  Bilateral values and Variability in TDC values

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Southeastern University, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided